CLINICAL TRIAL: NCT07170306
Title: A Study on the Prevalence and Clinical Characteristics of Cardiac Amyloidosis in Patients With Aortic Stenosis
Brief Title: Cardiac Amyloidosis in Patients With Aortic Stenosis
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CA-TAVR
Record Dates: First submitted 2025-09-05; First posted 2025-09-12 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Aortic Stenosis; Transthyretin Amyloid Cardiomyopathy
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — On the morning of the day after admission, 4 mL of elbow venous blood was routinely collected. The supernatant was separated and aliquoted into 3 EP tubes (500 μL per tube), then stored in a -80°C refrigerator. Repeated freezing and thawing was avoided, and the samples were kept for subsequent analysis. Serum samples were thawed at room temperature for more than 30 minutes, and subsequent procedures were performed after complete thawing.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ATTR-AS group: Patients were grouped according to the presence or absence of ATTR, i.e., into the isolated AS group and the ATTR-AS group.
  Interventions: Procedure: transcatheter aortic valve replacement (TAVR)
- AS group: Patients were grouped according to the presence or absence of ATTR, i.e., into the isolated AS group and the ATTR-AS group.
  Interventions: Procedure: transcatheter aortic valve replacement (TAVR)

INTERVENTIONS:
Procedure: transcatheter aortic valve replacement (TAVR) — TAVR is a minimally invasive cardiac interventional procedure that delivers a compressed artificial aortic valve to the diseased aortic valve site via peripheral blood vessels (e.g., the femoral artery) or the apex of the heart through a catheter, releases and deploys the valve to replace the original diseased valve leaflets, thereby restoring normal valve function and treating severe aortic stenosis (AS).

SUMMARY:
This study intends to conduct a prospective observation to investigate the prevalence of cardiac amyloidosis (CA) in patients with aortic stenosis (AS), compare the clinical characteristics between patients with isolated AS and those with AS complicated by CA (CA-AS), and simultaneously explore the impact of transcatheter aortic valve replacement (TAVR) on serum transthyretin (TTR) levels in patients with AS complicated by transthyretin amyloidosis (ATTR-AS), as well as its influence on the treatment outcomes of patients with isolated AS and ATTR-AS.

DETAILED DESCRIPTION:
Amyloid infiltration involving the aortic valve may cause endothelial damage, which in turn accelerates calcification and leads to the development or exacerbation of aortic stenosis (AS). Previous studies have shown that the comorbidity rate of transthyretin amyloid cardiomyopathy (ATTR-CA) and AS ranges from 4.9% to 16%, and this rate is particularly notable in patients who have undergone transcatheter aortic valve replacement (TAVR).

Currently, although small-scale studies have explored the prognosis of patients with AS complicated by CA, some conclusions are contradictory and have limitations. The present study intends to conduct a prospective observational study: on one hand, to investigate the prevalence of CA in patients with AS and compare the clinical characteristics between patients with isolated AS and those with CA-complicated AS (CA-AS); on the other hand, to explore the impact of TAVR on serum transthyretin (TTR) levels in patients with ATTR-complicated AS (ATTR-AS), as well as its influence on the treatment outcomes of patients with isolated AS and ATTR-AS.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥ 65 years and ≤ 85 years;
* Patients with moderate-to-severe degenerative aortic stenosis (AS) who are hospitalized and scheduled to undergo transcatheter aortic valve replacement (TAVR);
* Patients who voluntarily sign the Informed Consent Form (ICF) and are able to comply with the study-specified treatment plan, follow-up visits, laboratory tests, and other requirements.

Exclusion Criteria:

* Aortic stenosis (AS) caused by congenital diseases or rheumatic immune diseases;
* Severe renal impairment, chronic dialysis, or unresolved acute kidney injury after transcatheter aortic valve replacement (TAVR);
* Terminal-stage diseases with an expected life span of < 6 months;
* Participation in other ongoing investigational studies of drugs or medical devices that have not yet been completed;
* Patients who are unable to attend the follow-up visits scheduled in the study;
* Failure to undergo TAVR surgery, transfer to surgical treatment, or in-hospital death.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients admitted to the Cardiology Ward who undergo transcatheter aortic valve replacement (TAVR) for severe aortic stenosis (AS) from May 2025 to May 2028.
Sampling Method: Non-Probability Sample
Enrollment: 143 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality Composite endpoint of death and first hospitalization for heart failure In accordance with | baseline, 1 month, 3 months, 6 months, and 12 months
  All-cause mortality is a statistical measure that counts all deaths in a specific population over a given time period, regardless of the cause of death.
Composite endpoint of death and first hospitalization for heart failure | 12 months
  In accordance with the Valve Academic Research Consortium-2 (VARC-2) criteria, the composite endpoints for early safety and clinical efficacy after transcatheter aortic valve replacement (TAVR) were evaluated.
Change in serum transthyretin (TTR) level from baseline | baseline, 1 month, 3 months, 6 months, and 12 months
  At baseline, 1 month, 3 months, 6 months, 12 months, the serum TTR levels were measured to assess the changes compared to the baseline.

SECONDARY OUTCOMES:
Change in N-terminal pro-B-type natriuretic peptide (NT-proBNP) level from baseline | baseline, 1 month, 3 months, 6 months, and 12 months
  NT-proBNP levels were measured at baseline, 1 month, 3 months, 6 months, and 12 months, and the change from baseline was evaluated.
Change in New York Heart Association (NYHA) functional classification from baseline | baseline, 1 month, 3 months, 6 months, and 12 months
  NYHA functional classification was assessed at baseline, 1 month, 3 months, 6 months, and 12 months, and the change from baseline was evaluated. The assessment was based on the New York Heart Association Functional Classification Scale, which is a 4-level ordinal scale with a minimum value of Class Ⅰ and a maximum value of Class Ⅳ. For this scale, higher scores represent worse clinical outcomes:
  Class Ⅰ: No limitation of physical activity Class Ⅱ: Slight limitation of physical activity Class Ⅲ: Marked limitation of physical activity Class Ⅳ: Unable to carry on any physical activity without symptoms
Change in quality of life from baseline | baseline, 6 months, and 12 months
  In this study, the Minnesota Living With Heart Failure Questionnaire (MLHFQ) was used to assess patients' quality of life at baseline, 6 months, and 12 months. The MLHFQ corresponds to the full name Minnesota Living With Heart Failure Questionnaire, a disease-specific tool for evaluating heart failure-related quality of life. This scale has a total score range of 0 (minimum) to 105 (maximum). A higher total score reflects more severe quality of life impairment (i.e., worse outcome), while a lower score indicates better physical and psychological well-being in patients with heart failure.
Change in Left Ventricular Ejection Fraction (LVEF) from baseline | baseline, 1 month, 3 months, 6 months, and 12 months
  LVEF changes were evaluated at baseline, 1 month, 3 months, 6 months, and 12 months.

OTHER OUTCOMES:
Ventricular remodeling indices | at baseline and 12 months
  Cardiac Magnetic Resonance (CMR) was used to assess patients' ventricular function and structure at baseline and 12 months.
Echocardiographic indices | baseline, 1 month, 3 months, 6 months, and 12 months
  Echocardiography was used to assess ventricular systolic function at baseline, 1 month, 3 months, 6 months, and 12 months.
Change in cardiac troponin T (cTnT) level from baseline | baseline, 1 month, 3 months, 6 months, and 12 months
  The change in cTnT level from baseline was evaluated at baseline, 1 month, 3 months, 6 months, and 12 months.
99Tcm-phosphonate (99Tcm-PYP) bone scan indices | baseline, 12 months
  Patients underwent 99Tcm-PYP bone scans at baseline and 12 months, and the visual scoring grades and heart/contralateral lung (H/CL) ratios were recorded.
Incidence of postprocedural complications | 1 month
  Incidence of postprocedural complications, such as acute kidney injury, major bleeding, vascular complications, stroke, and new pacemaker implantation.
Number of participants with adverse events (AEs) and serious adverse events (SAEs) within 12 months | 12 months
  Number of participants with one or more AEs and SAEs within 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Daxin Zhou, Principal Investigator — Fudan University

IPD SHARING:
Plan to Share IPD: No